CLINICAL TRIAL: NCT01085409
Title: The Q in the QALY: Exploring New Methods
Brief Title: The Q in the Quality Adjusted Life Years (QALY): Exploring New Methods
Acronym: MOMENTUM
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Adelante, Centre of Expertise in Rehabilitation and Audiology (Other)
Responsible Party: Principal Investigator, Iris Maes, MSc, Maastricht University Medical Center
Other Study IDs: 80-82500-98-9207
Record Dates: First submitted 2010-03-10; First posted 2010-03-11 (Estimated); Last update posted 2013-05-07 (Estimated); Status verified 2013-05

CONDITIONS: Healthy
Keywords: experienced utility; decision utility; subjective well-being; experience sampling method; day reconstruction method; Quality of life

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Tinnitus: Patients with tinnitus
- Artery disease: Subjects with mobility constraints as a results of severe artery disease which in some cases led to leg amputation.
- Anxiety: Subjects with anxiety complaints
- Controls: Healthy controls

SUMMARY:
Aim: The aim of this proposal is to investigate the potential use and value of experienced utility, as measured by the Experience Sampling Method and the Day Reconstruction Method, in the economic evaluation of health care.

Methods: Three samples of 46 patients with different conditions one sample of 46 healthy controls will be included in the study. The Experience Sampling Method (ESM) and the Day Reconstruction Method (DRM) will be adapted and subsequently used to measure experienced utility. Decision utilities will be elicited by traditional preference based methods.

Expected results: The expected results of this study are threefold. First, unified versions of the ESM and DRM for use in the economic evaluation of health care will be developed and applied. Second, a rich dataset will allow us to investigate the differences between the results of experienced utilities derived from these methods, with the traditional preference based measures. Third, the normative implications of the use of QALYs based on either decision utilities, experienced utilities, or a combination of the two, for health care resource allocation decisions, will be examined.

Keywords: experienced utility, decision utility, subjective well-being, experience sampling method, day reconstruction method

DETAILED DESCRIPTION:
This study explores new methodology regarding the measurement of health state utilities. A new pharmaceutical is nowadays only reimbursed if there is evidence of cost-effectiveness. This can be determined by different types of economic evaluations, of which cost-utility analysis (CUA) is preferred in most guidelines. In CUA the health outcome of a technology is measured in quality adjusted life years (QALY). Utilities to calculate QALYs should be based on decisions under uncertainty (decision utilities). However, the health care literature describes several problems that lead to bias in the measurement of decision utilities. These biases lead to an inaccurate estimation of the value of a health state and can therefore cause policy makers to allocate resources inefficiently. To solve some of these problems, it was suggested to determine experiences associated with different health states by measuring well-being moment-to-moment (experienced utility) by the Experience Sampling Method or the Day Reconstruction Method.

Differences between the utilities measured using traditional preference based measures (decision utility), and using the new state-of-art methods ESM and DRM (experienced utility) in a range of populations with differing conditions and severity of health state will be investigated. Since somatic, psychosomatic and psychological conditions are likely to differ in the way they experience and affect well-being, we will involve patient groups from each category in this study as well as healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Diagnose on one of the diseases under investigation
* 18 years or older

Exclusion Criteria:

* not being able to read in Dutch
* not able to handle the ESM device because of impaired motor skills

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from the Maastricht University Medical Hospital or Adelante centre of expertise in rehabilitation and audiology. Healthy controls will be recruited by advertisement in local newspapers and flyers.
Sampling Method: Non-Probability Sample
Enrollment: 139 (Actual)
Dates: Start 2010-04; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Quality of Life | During 1 week
  The primary outcome measure of this study is quality of life as measured with a Visual Analogue Scale (VAS), the EuroQol, the Experience Sampling Method, the Day Reconstruction Method and the Time trade-off.

SECONDARY OUTCOMES:
Life satisfaction | 2 times
  Life satisfaction as mesured with te Satisfaction with Life Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Iris Maes, MSc, Principal Investigator — Maastricht Universitair Medical Centre; Manuela Joore, PhD, Principal Investigator — Maastricht University Medical Centre
Locations (2):
- Netherlands (2):
  - Adelante, Hoensbroek, Limburg
  - Maastricht University Medical Hospital, Maastricht, Limburg